CLINICAL TRIAL: NCT02568423
Title: A Single-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of LY3074828 in Japanese and Caucasian Healthy Subjects
Brief Title: A Study of Mirikizumab (LY3074828) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16172; I6T-JE-AMAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mirikizumab IV (Experimental): Participants received 200mg Mirikizumab by intravenously.
  Interventions: Drug: Mirikizumab - IV
- Mirikizumab SC (Experimental): Participants received single dose of either 60mgor 200mg 0r 600mg or 1200mg or 2400mg Mirikizumab by subcutaneously.
  Interventions: Drug: Mirikizumab - SC
- Placebo IV (Placebo Comparator): Participants received placebo by intravenously.
  Interventions: Drug: Placebo - IV
- Placebo SC (Placebo Comparator): Participants received placebo by subcutaneously.
  Interventions: Drug: Placebo - SC

INTERVENTIONS:
Drug: Mirikizumab - IV — Administered IV
  Other Names: LY3074828
  Arms: Mirikizumab IV
Drug: Mirikizumab - SC — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab SC
Drug: Placebo - IV — Administered IV
  Arms: Placebo IV
Drug: Placebo - SC — Administered SC
  Arms: Placebo SC

SUMMARY:
The main purpose of this study is to explore the safety and tolerability of mirikizumab in healthy Japanese and Caucasian participants. The study will also estimate how much mirikizumab gets into the blood stream and how long it takes the body to remove it. The study is expected to last about 16 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination.
* Are first generation Japanese or are Caucasian.
* Have a body mass index (BMI) of 18.0 kilograms per square meter (kg/m2) to 32.0 kg/m2, inclusive, at screening.
* Have a body weight of 40.0 kg or higher for Cohorts 1, 2, 3 and 4, and 48.0 kg or higher for Cohort 5 and 6.

Exclusion Criteria:

* Have had symptomatic herpes zoster within 3 months of screening.
* Show evidence of active or latent tuberculosis (TB), as documented by medical history and examination, chest x-rays (posterior anterior and lateral), and TB testing.
* Have received live vaccine(s) within 1 month of screening or intend to during the study.
* Are immunocompromised.
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- WCCT Global, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Subcutaneous (SC): Participants received placebo subcutaneously (SC).
- Placebo IV: Participants received placebo by IV.
- 60mg Mirikizumab IV: Participants received 60mg Mirikizumab by IV.
- 200mg Mirikizumab SC: Participants received 200mg Mirikizumab by SC.
- 200mg Mirikizumab IV: Participants received 200mg Mirikizumab by IV.
- 600mg Mirikizumab IV: Participants received 600mg Mirikizumab by IV.
- 1200mg Mirikizumab IV: Participants received 1200mg Mirikizumab by IV.
- 2400mg Mirikizumab IV: Participants received 2400mg Mirikizumab by IV.
Period: Overall Study
Arm/Group | Placebo Subcutaneous (SC) | Placebo IV | 60mg Mirikizumab IV | 200mg Mirikizumab SC | 200mg Mirikizumab IV | 600mg Mirikizumab IV | 1200mg Mirikizumab IV | 2400mg Mirikizumab IV
Started | 2 | 10 | 6 | 6 | 6 | 9 | 6 | 6
Received at Least One Dose of Study Drug | 2 | 10 | 6 | 6 | 6 | 9 | 6 | 6
Completed | 2 | 8 | 6 | 6 | 6 | 8 | 6 | 6
Not Completed | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo SC: Participants received placebo by SC.
- Total: Total of all reporting groups
Arm/Group | Placebo SC | Placebo IV | 60mg Mirikizumab IV | 200mg Mirikizumab SC | 200mg Mirikizumab IV | 600mg Mirikizumab IV | 1200mg Mirikizumab IV | 2400mg Mirikizumab IV | Total
Number analyzed (Participants) | 2 | 10 | 6 | 6 | 6 | 9 | 6 | 6 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (2.1) | 45.7 (10.6) | 49.3 (9.4) | 37.3 (8.8) | 41.7 (16.0) | 46.8 (11.9) | 37.8 (11.9) | 45.2 (6.0) | 44 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 3 | 3 | 5 | 5 | 3 | 5 | 31
  Male | 1 | 4 | 3 | 3 | 1 | 4 | 3 | 1 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 3 | 0 | 2 | 2 | 1 | 9
  Not Hispanic or Latino | 2 | 9 | 6 | 3 | 6 | 7 | 4 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 3 | 3 | 3 | 5 | 3 | 3 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 5 | 3 | 3 | 3 | 4 | 3 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 10 | 6 | 6 | 6 | 9 | 6 | 6 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: SAE is any adverse event (AE) from this study that results in one of the following outcomes:
  1. death
  2. initial or prolonged inpatient hospitalization
  3. a life-threatening experience (that is, immediate risk of dying)
  4. persistent or significant disability/incapacity
  5. congenital anomaly/birth defect
  6. considered significant by the investigator for any other reason
Time Frame: Baseline through Day 85
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- 200mg Mirikizumab IV: Participants received 200mg Mirikizumab b IV.
Arm/Group | Placebo SC | Placebo IV | 60mg Mirikizumab IV | 200mg Mirikizumab IV | 200mg Mirikizumab SC | 600mg Mirikizumab IV | 1200mg Mirikizumab IV | 2400mg Mirikizumab IV
Number analyzed (Participants) | 2 | 10 | 6 | 6 | 6 | 9 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Mirikizumab.
Time Frame: Day 1: 0 (pre dose), end of infusion, 2, 6, 24, 72, 168, 240, 336, 504, 672, 1008, 1344, 1680, 2016 hr post dose for IV administration; Day 1: 0 (pre dose), 6, 24, 72, 168, 240, 336, 504, 672, 1008, 1344, 1680, 2016 hr post dose for SC administration
Population: All randomized participants who received at least one dose of Mirikizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per Milliliter (μg/mL)
Arm/Group | 60mg Mirikizumab IV | 200mg Mirikizumab SC | 200mg Mirikizumab IV | 600mg Mirikizumab IV | 1200mg Mirikizumab IV | 2400mg Mirikizumab IV
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 6 | 6
Microgram per Milliliter (μg/mL) | 23.1 (9) | 11.8 (39) | 78.8 (13) | 250 (16) | 454 (11) | 985 (20)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration (AUC) Curve From Time Zero to Infinity of Mirikizumab
Description: Pharmacokinetics: Area Under the Concentration (AUC) Curve from Time Zero to Infinity of Mirikizumab.
Time Frame: as for outcome 2
Population: All randomized participants who received at least one dose of Mirikizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram day per milliliter (μg*day/mL)
Arm/Group | 60mg Mirikizumab IV | 200mg Mirikizumab SC | 200mg Mirikizumab IV | 600mg Mirikizumab IV | 1200mg Mirikizumab IV | 2400mg Mirikizumab IV
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 6 | 6
Microgram day per milliliter (μg*day/mL) | 148 (29) | 210 (29) | 539 (12) | 1970 (24) | 2900 (14) | 5990 (12)

ADVERSE EVENTS:
Time Frame: Up to 88 days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo SC | Placebo IV | 60mg Mirikizumab IV | 200mg Mirikizumab SC | 200mg Mirikizumab IV | 600mg Mirikizumab IV | 1200mg Mirikizumab IV | 2400mg Mirikizumab IV
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/10 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/10 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/2 | 5/10 | 3/6 | 1/6 | 2/6 | 1/9 | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC (N=2) | Placebo IV (N=10) | 60mg Mirikizumab IV (N=6) | 200mg Mirikizumab SC (N=6) | 200mg Mirikizumab IV (N=6) | 600mg Mirikizumab IV (N=9) | 1200mg Mirikizumab IV (N=6) | 2400mg Mirikizumab IV (N=6)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT02568423/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT02568423/SAP_001.pdf